CLINICAL TRIAL: NCT01731652
Title: Phase II Pilot Study With TMX 101 in Patients With Carcinoma In Situ (CIS) Bladder Cancer
Brief Title: Study With TMX-101 in Patients With Carcinoma In Situ (CIS) Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telormedix SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMX-101-003
Record Dates: First submitted 2012-11-12; First posted 2012-11-22 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Carcinoma in Situ; Non Muscle Invasive Bladder Cancer
Keywords: bladder cancer; carcinoma in situ; non muscle invasive bladder cancer
MeSH Terms: conditions — Carcinoma in Situ; Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMX-101 (Experimental): TMX-101 0.4% (200 mg in 50 ml) instilled in the bladder once weekly for 6 weeks
  Interventions: Drug: TMX-101

INTERVENTIONS:
Drug: TMX-101
  Other Names: Imiquimod

SUMMARY:
This is a Phase II pilot study to explore the effect of intravesical TMX-101 in patients with CIS bladder cancer, as assessed by histology and cytology after TMX-101 treatment.

DETAILED DESCRIPTION:
This study is an open label, pilot study of TMX-101 in the treatment of carcinoma in situ. TMX-101 is a new formulation of Imiquimod optimized for intravesical delivery. Imiquimod possesses immune-stimulatory properties. TMX-101 is being developed as a potential treatment for patients with non-invasive bladder cancer, including patients with CIS bladder cancer.

Following confirmation of CIS by histology, patients will receive weekly instillations of TMX-101 for 6 weeks. Five to seven weeks after the last instillation, biopsies and cytology will be performed. Response to treatment will be determined based on cytology and tissue sample histology findings.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female patient is aged ≥18 years.
2. Pathologically-proven, recurrent, primary, secondary or concomitant carcinoma in situ disease, defined by having either Ta or T1 with CIS, or CIS alone. In cases with T1 tumor lesions, muscularis propria tissue should be in the resected specimen to confirm that it is tumor-free.
3. Patient has undergone mapping of the bladder between Days -28 and -14, with at least one biopsy providing pathological confirmation of CIS of the bladder. Slides must be available for a central pathology review.
4. Patient has undergone bladder washing for cytology between Days -28 and -1. In patients in whom Ta or T1 lesion(s) were resected, the bladder washing must have occurred after the resection. Slides must be available for a central cytology review.
5. Patient has an ECOG performance status 0-2.
6. Patient has adequate bone marrow, hepatic, and renal function within 4 weeks before Day 0.
7. Patient has read and understood the informed consent form and is willing and able to give informed consent.
8. Patient fully understands the requirements of the study and is willing to comply with all study visits and assessments.
9. If a woman of childbearing potential (WCBP), patient has a negative blood pregnancy test at the Screening visit. For the purposes of this study, WCBP is defined as a post-pubescent female, unless post-menopausal for at least 2 years, surgically sterile, or sexually inactive.
10. If patient is a WCPB or male patient with a female partner of childbearing potential, must be willing to avoid pregnancy by using an adequate method of contraception from 2 weeks before through 4 weeks after the last study drug treatment. Adequate contraception is defined as follows: 2 barrier methods or 1 barrier method with a spermicide or intrauterine device.

Exclusion Criteria:

1. Patient has evidence of muscle-invasive disease (i.e., T2 or higher)
2. In the Investigator's opinion, patient is not able to hold instillation for at least 1 hour.
3. In the Investigator's opinion, patient cannot tolerate intravesical administration or intravesical surgical manipulation.
4. Patient has received radiation therapy of pelvis within 12 months before the first study drug treatment.
5. Patient requires perioperative intravesical chemotherapy.
6. Patient has a history of malignancy of the upper urinary tract.
7. Patient has bone marrow impairment as evidenced by:

   * Hemoglobin <9.0 g/dL
   * Absolute neutrophil count (ANC) <1.5×109/L
   * Platelet count <120×109/L.
8. Patient has renal impairment, as evidenced by:

   * Serum creatinine >2× the upper limit of normal (ULN), and/or
   * Calculated creatinine clearance <40 mL/min.
9. Patient has liver function abnormality, as evidenced by:

   * Total bilirubin >1.5×ULN, or
   * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) >2.5×ULN.
10. Patient has a bleeding disorder, as evidenced by an international normalized ratio (INR) >1.5×ULN.
11. Patient is known to be positive for human immunodeficiency virus (HIV) or has active hepatitis B or C infection.
12. Patient has a clinically significant active infection at the time of the first study drug treatment.
13. Patient has any medical or psychiatric condition that, in the Investigator's opinion, might impair the patient's well-being or preclude adherence to the protocol or completing the study as per protocol.
14. Patient has suspected hypersensitivity to imidazoquinoline compounds, poloxamer 407, hydroxy propyl betacyclodextrin, or lactic acid.
15. If female, patient is pregnant or breast feeding.
16. Patient participated in any other protocol involving administration of an investigational agent within 3 months before Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To assess the activity of TMX-101, as determined by the number of patients who experience complete response (CR). | 5 to 7 weeks after the last TMX -101 instillation

SECONDARY OUTCOMES:
Proportion of patients experiencing adverse events (AEs), including serious adverse events (SAEs) and AEs leading to discontinuation from the study. | Patients will be followed through treatment and follow-up, for an expected total period of up to 13 weeks.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - BCG Oncology, Phoenix, Arizona
  - The Urology Center of Colorado, Denver, Colorado
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

REFERENCES:
- [Derived] Donin NM, Chamie K, Lenis AT, Pantuck AJ, Reddy M, Kivlin D, Holldack J, Pozzi R, Hakim G, Karsh LI, Lamm DL, Belkoff LH, Belldegrun AS, Holden S, Shore N. A phase 2 study of TMX-101, intravesical imiquimod, for the treatment of carcinoma in situ bladder cancer. Urol Oncol. 2017 Feb;35(2):39.e1-39.e7. doi: 10.1016/j.urolonc.2016.09.006. Epub 2016 Oct 26. PMID 28341495